CLINICAL TRIAL: NCT03798067
Title: Correlation Between Monitoring Renal Hemodynamics by Esophageal Ultrasound and Acute Kidney Injury After Heart Surgery.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Principal Investigator, Xuzhou Medical University
Other Study IDs: XYFY-2018-0008
Record Dates: First submitted 2019-01-01; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Creatinine, eGFR: blood was collected preoperatively, 4h postoperatively, and at least 3 days postoperatively in the morning.
  TIMP-2,IGPBP-7:Urine samples were collected before and after surgery at 4, 12 and 24 hours
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a common complication of cardiac surgery, which seriously affects the postoperative complication rate and mortality of patients.Acute kidney injury occurs in 5-30% of patients after cardiac surgery, but severe acute kidney injury requiring dialysis is relatively rare.At present, the diagnosis of AKI is based on serum creatinine (Scr) or urine volume. However, the changes of serum creatinine value have hysteresis, and the increase of serum creatinine level lags behind kidney injury for 48 ~ 72 h.Some drugs can also affect creatinine levels.Urine volume is also affected by many factors.Due to the lack of sensitivity and specificity of SCr, it is very important to find and adopt new early AKI markers.Kidney is an important metabolic organ of human body. Different from cerebrovascular system, kidney lacks automatic regulation ability and is easily affected by perfusion flow.Previous experiments have shown that placing a multi-plane esophageal probe into the human stomach through the esophagus can monitor the changes of left renal blood flow before, during and after cardiovascular surgery extracorporeal circulation, and has good repeatability, which may become an effective means to monitor renal blood flow during cardiovascular surgery.

In conclusion, this study intends to use esophageal ultrasound as a means to monitor renal blood flow, observe the changes of intraoperative renal hemodynamic indexes, and use KDIGO ( Kidney Disease:Improving Global Outcomes)as the standard of renal injury to explore the correlation between intraoperative hemodynamic changes and postoperative AKI, providing a new perspective for the pathophysiological study of AKI after cardiopulmonary bypass.

DETAILED DESCRIPTION:
The mechanism of acute kidney injury after CPB has not been fully elucidated, and current studies suggest that the main mechanisms are as follows:

(1) endogenous/exogenous nephrotoxic substances;(2) metabolic factors: mainly reflected in the preoperative status of patients, such as obesity, low body weight, etc.;(3) hemodynamic factors: hemodynamic instability is an important mechanism for further renal injury process such as ischemia reperfusion, which is mainly reflected in: a.preoperative and postoperative hypotension: cardiogenic shock caused by cardiac insufficiency and low cardiac displacement;Non-cardiogenic shock (vasoactive drugs/allergies/postoperative bleeding);b. hemodynamic instability of intraoperative intervention: deep anesthesia, intraoperative blood loss, CPB-related intraoperative low perfusion (long CPB time, low circulation flow, low mean arterial pressure in CPB), embolic release (atherosclerotic emboli/air emboli), aorta and distal arteriotomy;(4) neurohumoral system factors: hormones such as epinephrine, norepinephrine, renin and thyroxine change to varying degrees during cardiac surgery and CPB, thus affecting the body state and systemic blood vessels;(5) inflammation and oxidative stress.

Kidney is an important metabolic organ of human body. Different from cerebrovascular system, kidney lacks automatic regulation ability and is easily affected by perfusion flow.For patients at high risk of postoperative acute kidney injury, appropriate intraoperative perfusion may reduce the incidence of postoperative acute kidney injury.

Esophageal ultrasound was used as a means of monitoring renal blood flow to observe the changes in intraoperative renal hemodynamic indexes. Meanwhile, KDIGO was used as the standard for renal injury. AKI was divided into two groups according to whether postoperative AKI occurred, and the correlation between intraoperative hemodynamic changes and postoperative AKI in the two groups was discussed.It provides new ideas for the early diagnosis of postoperative acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70;
* Elective cardiopulmonary bypass for patients undergoing cardiac surgery

Exclusion Criteria:

* Acute myocardial infarction surgery within 7 days
* Emergency surgery
* Known renal artery stenosis, renal malformation;Renal failure
* Congenital esophageal malformation
* Patients with previous history of stomach and esophagus should avoid intraoperative esophageal ultrasound examination
* Existing acute kidney injury, kidney transplantation, chronic kidney disease and glomerular filtration rate less than 30 ml/min,
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients undergoing elective cardiac surgery in the Affiliated Hospital of Xuzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
AUC(RI) | RI monitored 30 minutes after cardiopulmonary bypass termination
  ROC curve（receiver operating characteristic curve）will be drawn according to the incidence of renal resistance index (RI) monitored by TEE and the incidence of postoperative AKI in patients, and AUC value(Area Under Curve) will be statistically analyzed.
AUC(PI) | PI monitored 30 minutes after cardiopulmonary bypass termination
  ROC curve will be drawn according to the incidence of renal pulsatility index (PI) monitored by TEE and the incidence of postoperative AKI in patients, and AUC value will be statistically analyzed.

SECONDARY OUTCOMES:
Changes in biomarkers | Before surgery and at 4 hours, 12 hours, and 24 hours after surgery
  Analysis of insulin-like growth factor-binding protein 7 (IGFBP7) and tissue inhibitor of metalloproteinases-2 (TIMP-2) concentrations (both induction factors for G1 cell cycle arrest are associated with acute kidney injury and are predicted as biomarkers).
Length of ICU stay | an average of 2 days
  All patients are routinely transferred to ICU after surgery
Length of hospital stay | an average of 10 days
  All patients are routinely transferred to ICU after surgery
Use of renal replacement therapy | Until 3 months after discharge
  The use of postoperative renal replacement therapy depends on the diagnosis and treatment of ICU staff.
Survival rate | At 1, 7 and 30 days after discharge
  Record the survival rate after hospital discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Dong Liu, M.S, Study Director — The Affiliated Hospital of Xuzhou Medical University

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data(IPD) will be available when this trial is finished and the article have been published.

REFERENCES:
- [Result] Weisse AB. Cardiac surgery: a century of progress. Tex Heart Inst J. 2011;38(5):486-90. PMID 22163121
- [Result] Wang Y, Bellomo R. Cardiac surgery-associated acute kidney injury: risk factors, pathophysiology and treatment. Nat Rev Nephrol. 2017 Nov;13(11):697-711. doi: 10.1038/nrneph.2017.119. Epub 2017 Sep 4. PMID 28869251
- [Result] Bellos I, Pergialiotis V, Kontzoglou K. Renal resistive index as predictor of acute kidney injury after major surgery: A systematic review and meta-analysis. J Crit Care. 2019 Apr;50:36-43. doi: 10.1016/j.jcrc.2018.11.001. Epub 2018 Nov 15. PMID 30471559
- [Result] Regolisti G, Maggiore U, Cademartiri C, Belli L, Gherli T, Cabassi A, Morabito S, Castellano G, Gesualdo L, Fiaccadori E. Renal resistive index by transesophageal and transparietal echo-doppler imaging for the prediction of acute kidney injury in patients undergoing major heart surgery. J Nephrol. 2017 Apr;30(2):243-253. doi: 10.1007/s40620-016-0289-2. Epub 2016 Mar 19. PMID 26995003